CLINICAL TRIAL: NCT05504720
Title: Pembrolizumab and Trastuzumab in Combination With FLOT in the Perioperative Treatment of HER2-positive, Localized Esophagogastric Adenocarcinoma - A Phase II Trial of the AIO Study Group - PHERFLOT -
Brief Title: Evaluating Pembrolizumab, Trastuzumab and FLOT as Perioperative Treatment of HER2-positive, Localized Esophagogastric Adenocarcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Organon Healthcare GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PHERFLOT; 2021-006512-87 (EudraCT Number); AIO-STO-0321 (Other: AIO-Studien GmbH)
Record Dates: First submitted 2022-08-15; First posted 2022-08-17 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Esophagogastric Adenocarcinoma
Keywords: gastric adenocarcinoma; GEJ adenocarcinoma; Her-2 positive esophagogastric adenocarcinoma
MeSH Terms: interventions — pembrolizumab; Trastuzumab; Ontruzant

STUDY DESIGN:
Intervention Model Description: All eligible patients will receive pembrolizumab at a dosage of 200 mg flat dose in combination with trastuzumab (6 mg/kg after loading dose of 8 mg/kg) every 3 weeks and 5-FU 2600 mg/m2 for 24 h, folinic acid 200 mg/m2, oxaliplatin 85 mg/m2 and docetaxel 50 mg/m2 (FLOT regimen) every 2 weeks for 8 weeks, followed by surgical resection 4 weeks after last preoperative treatment at the earliest, followed (within 4-10 weeks) by further 8 weeks of the same regime, followed by pembrolizumab 200 mg and trastuzumab 6 mg/kg alone for up to 11 cycles. In total 1 year of systemic treatment (17 pembrolizumab/ trastuzumab administrations max. per patient incl. pre- and postoperative chemo-immunotherapy).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pembrolizumab Trastuzumab (Experimental): Single arm with pembrolizumab (200 mg flat dose over 30 min IV) on day 1, 22 and 43 plus trastuzumab (loading dose 8 mg/kg IV over 90 min at day 1 and maintenance dose 6 mg/kg IV over 30 min) on day 22 and 43 plus FLOT in four 2-week treatment cycles prior to undergoing surgery. Following surgery, patients will receive four further 2-week cycles of pembrolizumab+trastuzumab + FLOT followed by pembrolizumab (200 mg flat dose) and trastuzumab (6 mg/kg) alone for up to 11 further cycles (Q3W).
  Interventions: Drug: Pembrolizumab; Drug: Trastuzumab; Drug: FLOT

INTERVENTIONS:
Drug: Pembrolizumab — 200 mg flat dose, IV, over 30 minutes; day 1, 22, 43 (8 weeks) pre- and post-surgery, followed by post chemotherapy phase day 1 q3w for 11 cycles; max. 17 applications
  Other Names: Keytruda
Drug: Trastuzumab — loading dose 8 mg/kg IV over 90 min: day 1 pre- and post-surgery; maintenance dose 6 mg/kg IV over 30 min: Day 22, 43 pre- and post-surgery; followed by 6 mg/kg post chemotherapy phase, day 1 q3w for 11 cycles; max. 17 applications
  Other Names: Ontruzant
Drug: FLOT — Docetaxel 50 mg/m² IV over 1 hour plus Oxaliplatin 85 mg/m² IV over 2 hours plus Folinic Acid 200 mg/m² IV over 1 hour plus 5-FU 2600 mg/m² IV over 24 hours every 2 weeks (day 1, 15, 29, 43) for 8 weeks pre- and 8 weeks post-surgery

SUMMARY:
The study is an open-label, single arm, multicenter phase II trial investigating the clinical activity of a perioperative therapy consisting of a combination of pembrolizumab, trastuzumab and FLOT, followed by pembrolizumab plus trastuzumab alone for a maximum systemic treatment duration of one year in patients with Her-2 positive localized esophagogastric adenocarcinoma.

DETAILED DESCRIPTION:
Her-2 positive patients suffering from localized esophagogastric adenocarcinoma (≥ T2 any N+ or any T N+) without evidence of metastatic disease will be included in the study. Eligible subjects will receive a combination of pembrolizumab and trastuzumab with FLOT 8 weeks pre- as well as post-surgery, followed by pembrolizumab and trastuzumab treatment for up to one year (maximum of 17 administrations of systemic treatment with pembrolizumab and trastuzumab incl. pre- and postoperative chemo-immunotherapy) or until tumor relapse/progression or occurrence of limiting toxicity.

The primary objective of this phase II study is to demonstrate the efficacy of the FLOT/trastuzumab/pembrolizumab regimen in terms of an improvement in disease free survival (DFS) according to RECIST v1.1 and an increase in the pathological complete response (pCR) rate compared to historical controls (interim read out after surgery of last patient in study with 18 months recruitment after 24 months). Secondary objectives are further efficacy and tolerability parameters, including overall response rate according to RECIST v1.1, R0 resection rate, overall survival, safety, and tolerability (including perioperative morbidity).

The exploratory objective is to assess whether clinical efficacy correlates with molecularly-defined subgroups (PD-L1 expression, MSI subtypes, and others).

30 patients will be enrolled in this trial.

ELIGIBILITY:
Inclusion Criteria:

1. The participant provides written informed consent for the trial.
2. Male/female* participants who are at least 18 years of age on the day of signing informed consent.

   *There are no data that indicate special gender distribution. Therefore, patients will be enrolled in the study gender-independently.
3. In the investigator's judgement, participant is willing and able to comply with the study protocol including the planned surgical treatment
4. Histologically confirmed adenocarcinoma of the GEJ (Type I-III according to Sievert´s classification) or the stomach (cT2, cT3, cT4, any N category, M0), or (any T, N+, M0) that:

   * is not infiltrating any adjacent organs or structures by CT or MRI evaluation
   * does not involve peritoneal carcinomatosis
   * is considered medically and technically resectable Note: the absence of distant metastases must be confirmed by CT or MRI of the thorax and abdomen, and, if there is clinical suspicion of osseous lesions, a bone scan. If peritoneal carcinomatosis is suspected clinically, its absence must be confirmed by laparoscopy. Diagnostic laparoscopy is mandatory in patients with T3 or T4 tumors of the diffuse type histology in the stomach.
5. Participants must have HER2-positive disease defined as either IHC 3+ or IHC 2+, the latter in combination with ISH+, as assessed locally by a certified test on primary tumor (see Appendix 4)
6. Participants must be candidates for potential curative resection as determined by the treating surgeon
7. No prior systemic-anti cancer therapy (e.g. cytotoxic or targeted agents or radiotherapy)
8. No prior partial or complete esophagogastric tumor resection
9. ECOG (Eastern Cooperative Oncology Group) performance status score of 0 or 1
10. Male participants: A male participant must agree to use a contraception as detailed in Appendix 2 of this protocol during the treatment period and for at least 6 months after the last dose of study intervention and refrain from donating sperm during this period.

    Female participants: A female participant is eligible to participate if she is not pregnant (see Appendix 2), not breastfeeding, and at least one of the following conditions applies:
    * Not a woman of childbearing potential (WOCBP) as defined in Appendix 2 OR
    * A WOCBP who agrees to follow the contraceptive guidance as given in Appendix 2 during the treatment period and for at least 7 months after the last dose of study intervention.
11. Participants have adequate organ function as defined in the following table (Table 2). Specimens must be collected within 14 days prior to enrolment (also to be repeated if older than 14 days at day of first treatment).

Hematological:

* Absolute neutrophil count (ANC) ≥ 1500/μL
* leucocytes ≥ 3000/μL
* Thrombocytes ≥ 100 000/μL
* Hemoglobin ≥ 9.0 g/dL or ≥ 5.6 mmol/L (Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within the last 2 weeks)

Renal:

• Measured or calculated (b) creatinine clearance≥ 50 mL/min

Hepatic:

* Total bilirubin ≤ 1.5 ×ULN OR direct bilirubin ≤ ULN for participants with total bilirubin levels > 1.5 × ULN
* AST (SGOT) and ALT (SGPT) ≤ 2.5 × ULN Coagulation
* International normalized ratio (INR) OR prothrombin time (PT) and
* Activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants ALT (SGPT)=alanine aminotransferase (serum glutamic pyruvic transaminase); AST (SGOT)=aspartate aminotransferase (serum glutamic oxaloacetic transaminase); GFR=glomerular filtration rate; ULN=upper limit of normal.

Exclusion Criteria:

1. Participants with involved retroperitoneal (e.g. para-aortal, paracaval or interaortocaval lymph nodes) or mesenterial lymph nodes (distant metastasis!)
2. A WOCBP who has a positive urine pregnancy test within 72 hours prior to start of study intervention (see Appendix 2). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
3. Received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX-40, CD137).
4. Participant received colony-stimulating factors (e.g. granulocyte colony-stimulating factor [G-CSF], granulocyte-macrophage colony-stimulating factor [GM-CSF] or recombinant erythropoietin) within 28 days prior to the first dose of study intervention.
5. Major surgery within 2 weeks of starting study intervention and patients must have recovered from any effects of any major surgery.
6. Concomitant use of drugs inhibiting (dihydropyrimidine dehydrogenase) DPD activity (including sorivudine, brivudine), the required wash out phase is 4 weeks before start of the study intervention.
7. Inadequate cardiac function (LVEF value < 55 %) as determined by echocardiography
8. Resting ECG indicating uncontrolled, potentially reversible cardiac conditions, as judged by the investigator (e.g., unstable ischemia, uncontrolled symptomatic arrhythmia, congestive heart failure, QTcF prolongation > 500 ms, electrolyte disturbances, etc.), or patients with congenital long QT syndrome.
9. Participant has received a live vaccine or live-attenuated vaccine within 30 days prior to the first dose of study drug. Administration of killed vaccines is allowed.
10. Participant is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention.
11. Participant has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
12. Participant has a known additional malignancy that is progressing or has required active treatment within the past 2 years. Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin or carcinoma in situ (e.g., breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
13. Participant has myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML) or with features suggestive of MDS/AML.
14. History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion protein; known hypersensitivity to Chinese hamster ovary cell products or to any component of the pembrolizumab or trastuzumab formulation
15. Any known contraindication (including hypersensitivity) to docetaxel, 5-FU, folinic acid/leucovorin, or oxaliplatin.
16. Known DPD deficiency. Patients with a reduced DPD activity (CPIC activity score of 1.0-1.5) might participate in the study and receive a reduced dosage of 5-FU after discussion with the coordinating investigator and sponsor [https://cpicpgx.org/guidelines/guideline-for-fluoropyrimidines-and-dpyd/]
17. Participant has active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
18. Participant has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
19. Participant has an active infection requiring systemic therapy.
20. Participant has a known history of Human Immunodeficiency Virus (HIV) infection
21. Participant has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA is detected) infection.
22. Participant is considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease on High Resolution Computed Tomography (HRCT) scan, previous allogenic bone marrow/blood transplantation or any psychiatric disorder or substance abuse that prohibits obtaining informed consent.
23. Participant is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 6 months after the last dose of study intervention.
24. Participant has had an allogenic tissue/solid organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2023-02-13 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival after 2 years co-primary endpoint | 2 years after enrolment
  Disease-free survival is defined as the proportion of patients being tumor/disease free and alive 2 years after enrolment.
Pathological complete response rate co-primary endpoint | after surgery, i.e. approx. 12 weeks after enrolment
  The pCR rate is defined as the absence of residual tumor based on evaluation of the resected esophagogastric specimen in the primary tumor by local pathology.

SECONDARY OUTCOMES:
Overall response rate (ORR) | up to 1 year after enrolment
  Overall response rate, defined as percentage of patients with CR and PR according to RECIST v1.1
Overall survival (OS) | up to 52 months
  Overall survival is defined as time from enrolment to the date of death of any cause. If no event is observed (e.g., lost to follow-up) OS is censored at the date of last subject contact. Subjects who are alive will be censored at the last known alive dates.
R0 resection rate | after surgery, i.e. approx. 12 weeks after enrolment
  R0 resection is defined as a microscopically margin negative resection with no gross or microscopic tumor remains in the areas of the primary tumor and/or sampled regional lymph nodes based on evaluation by the local pathologist
Feasibility rate | up to 32 weeks
  Feasibility rate - severe toxicity/withdrawal rate before the last postoperative administration of pembrolizumab/trastuzumab/FLOT has been completed.
Incidence and severity of adverse events according to CTC criteria | up to 18 months (max. 1 year treatment plus 90 days after last treatment)
  (Serious) adverse events - recorded and graded according to NCI-CTCAE V5.0. Occurrence of (serious) adverse events at any time during the study. Description by nature (System Organ Class and Preferred Term), severity and causal relationship to drug administration.

CONTACTS AND LOCATIONS:
Overall Officials: Salah Al-Batran, Prof. Dr., Study Director — Institut für Klinische Krebsforschung IKF GmbH
Locations (13):
- Germany (13):
  - Charité - Universitätsmedizin Berlin / Campus Virchow Klinikum (CVK), Berlin
  - MVZ Onkologischer Schwerpunkt, Berlin
  - KEM | Klinik für Internistische Onkologie gGmbH, Essen
  - Institut für Klinisch-Onkologische Forschung am Krankenhaus Nordwest, Frankfurt am Main
  - Hämatologisch-Onkologische Praxis Eppendorf, Hamburg
  - Nationales Centrum für Tumorerkrankungen, Heidelberg
  - St. Anna Hospital Herne, Herne
  - Tagestherapiezentrum (TTZ) am Interdisziplinären Tumorzentrum (ITM), Mannheim
  - Klinikum rechts der Isar der TU München, München
  - Klinikum Nürnberg, Nuremberg
  - Krankenhaus Barmherzige Brüder, Regensburg
  - Universitätsklinikum Ulm, Ulm
  - Klinikum Wolfsburg, Wolfsburg

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared.

REFERENCES:
- [Derived] Stein A, Goekkurt E, Al-Batran SE, Moosmann N, Ettrich TJ, Goetze T, Gruen B, Homann N, Lorenzen S, Hofheinz RD, Rempel V, Siegler G, Muller C, Thiele B, Broering T, Cruz MS, Pauligk C, Binder M, Tintelnot J. Perioperative pembrolizumab, trastuzumab and FLOT in HER2-positive localized esophagogastric adenocarcinoma: a phase 2 trial. Nat Med. 2025 Dec;31(12):4197-4204. doi: 10.1038/s41591-025-03979-y. Epub 2025 Oct 18. PMID 41109919
- [Derived] Tintelnot J, Stein A, Al-Batran SE, Ettrich T, Gotze T, Grun B, Haag GM, Heuer V, Hofheinz RD, Homann N, Broring TS, Cruz MS, Kurreck A, Lorenzen S, Moosmann N, Muller C, Schuler M, Siegler G, Binder M, Gokkurt E. Pembrolizumab and trastuzumab in combination with FLOT in the perioperative treatment of HER2-positive, localized esophagogastric adenocarcinoma-a phase II trial of the AIO study group (AIO STO 0321). Front Oncol. 2023 Oct 16;13:1272175. doi: 10.3389/fonc.2023.1272175. eCollection 2023. PMID 37909020